CLINICAL TRIAL: NCT04268927
Title: Extended Letrozole Regimen Co-treatment With Gonadotropin Releasing Hormone Antagonist Protocol Versus Gonadotropin Releasing Hormone Antagonist Protocol in Poor Responders Undergoing IVF-ET. A Randomized Controlled Trial
Brief Title: Extended Letrozole Regimen Co-treatment With Gonadotropin Releasing Hormone Antagonist Protocol Versus Gonadotropin Releasing Hormone Antagonist Protocol in Poor Responders Undergoing IVF-ET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: letrozole/ GnRH ant
Record Dates: First submitted 2020-02-12; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Infertility
Keywords: Letrozole ,IVF, poor responders , GnRH antagonist
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH ant/letrozole (Experimental): Letrozole (Femara; Novertis pharma AG, Basle, Switzerland) is administered starting on cycle day one for 8 consecutive days . The dose of letrozole is 5mg /day during the first 5 days of cycle and 2.5 mg/day during the subsequent 3 days .
  Highly purified urinary FSH (HP-uFSH) (Fostimon, IBSA) 300 IU/day is started on cycle day 5 and is continued until and including the day of HCG administration. Starting from cycle day 8 , the dose of HP-uFSH is adjusted individually according to ovarian response which is monitored using transvaginal ultrasound and serum estradiol.
  GnRH antagonist (cetrorelix acetate)(Cetrotide®) 0.25 mg S.C once daily is started when the leading follicle is 14 mm in mean diameter and is continued until and including the day of HCG administration .
  Interventions: Drug: GnRH ant/letrozole
- GnRH ant (Active Comparator): Highly purified urinary FSH (HP-uFSH) (Fostimon, IBSA) 300 IU/day is started on cycle day 5 and is continued until and including the day of HCG administration. Starting from cycle day 8 , the dose of HP-uFSH is adjusted individually according to ovarian response which is monitored using transvaginal ultrasound and serum estradiol.
  GnRH antagonist (cetrorelix acetate)(Cetrotide®) 0.25 mg S.C once daily is started when the leading follicle is 14 mm in mean diameter and is continued until and including the day of HCG administration .
  Interventions: Drug: GnRH ant

INTERVENTIONS:
Drug: GnRH ant/letrozole — Letrozole (Femara; Novertis pharma AG, Basle, Switzerland) is administered starting on cycle day one for 8 consecutive days . The dose of letrozole is 5mg /day during the first 5 days of cycle and 2.5 mg/day during the subsequent 3 days .
  Highly purified urinary FSH (HP-uFSH) (Fostimon, IBSA) 300 IU/day is started on cycle day 5 and is continued until and including the day of HCG administration. Starting from cycle day 8 , the dose of HP-uFSH is adjusted individually according to ovarian response which is monitored using transvaginal ultrasound and serum estradiol.
  GnRH antagonist (cetrorelix acetate)(Cetrotide®) 0.25 mg S.C once daily is started when the leading follicle is 14 mm in mean diameter and is continued until and including the day of HCG administration .
  Arms: GnRH ant/letrozole
Drug: GnRH ant — Highly purified urinary FSH (HP-uFSH) (Fostimon, IBSA) 300 IU/day is started on cycle day 5 and is continued until and including the day of HCG administration. Starting from cycle day 8 , the dose of HP-uFSH is adjusted individually according to ovarian response which is monitored using transvaginal ultrasound and serum estradiol.
  GnRH antagonist (cetrorelix acetate)(Cetrotide®) 0.25 mg S.C once daily is started when the leading follicle is 14 mm in mean diameter and is continued until and including the day of HCG administration .
  Arms: GnRH ant

SUMMARY:
The object of this study is to evaluate the efficacy of extended letrozole co-treatment with GnRH-antagonist protocol in ovarian stimulation of poor responder patients undergoing IVF-ET.

DETAILED DESCRIPTION:
Poor response to controlled ovarian stimulation (COH) is estimated to occur in 9-24 % of all IVF cycles. Although there is no consensus on the definition of poor response to COH, inability to produce adequate number of mature follicles( ≤ 2-5) or to recruit adequate number of oocytes ( ≤ 3 oocytes ) in response to standard stimulation protocols are the main criteria used for diagnosis of poor responders .

Patients with poor response to COH usually have higher cyclical cancelation rate , poor embryo quality and less number of embryos suitable for transfer or cryopreservation .

During the past decade gonadotropin releasing hormone antagonists (GnRHant) were widely used in the treatment of patients with poor response to standard gonadotropin releasing hormone agonist (GnRHa) protocols .In contrast to GnRHa, GnRHant is administered at the late follicular phase and therefore don't suppress the early follicular phase endogenous gonadotropins and has no suppressive effect on ovarian function at the stage of follicular recruitment.Several studies comparing GnRHant protocol with the standard GnRHa long protocol revealed a reduction in the duration of stimulation , dose of required gonadotropins , and the costs of IVF cycle with GnRHant as well as equivalent pregnancy rates .

In 2001, Mitwally and Casper introduced letrozole ( a third generation non steroidal aromatase inhibitor licensed for treatment of hormonally-responsive breast cancer after surgery ) as new ovulation induction agent in clomiphene citrate resistant patients with polycystic ovary syndrome (PCOS) . Subsequent studies confirmed the effectiveness of letrozole in induction of ovulation in women with PCOS and in superovulation (either alone or in combination with gonadotropins ) .

In patients with poor response undergoing IVF, several studies revealed that the combination of letrozole ( 2.5 mg or 5 mg/day for 5 consecutive days in early follicular phase ) with GnRHant protocol improved the ovarian response and reduced the gonadotrophin dose required. On the other hand , Schoolcraft et al reported that letrozole(2.5 mg/day from cycle day 3 to 7)/GnRHant protocol has no advantages over microdose flare GnRHa protocol.

The ideal dose and duration of letrozole administration for ovulation and superovulation is still not clear. Several studies comparing two doses of letrozole (2.5 mg or 5 mg) in superovulation suggested that the higher dose might be associated with more follicles developing.

In almost all studies to date , letrozole was administered for five consecutive days in early follicular phase . In only one study , letrozole (2.5 mg/day) was administered for ten consecutive days starting on day 1 of menstrual cycle . In that study , prolonged administration of letrozole produced more mature follicles and pregnancies than short letrozole therapy regimen in patients with clomiphene citrate resistant polycystic ovary syndrome .

The investigators designed this randomized controlled trial to evaluate the efficacy of extended letrozole co-treatment with GnRH-antagonist protocol in ovarian stimulation of poor responder patients undergoing IVF-ET

ELIGIBILITY:
Inclusion Criteria:

* Poor responders according to the ESHRE Bologna criteria

Exclusion Criteria:

Age > 42 years FSH> 12 IU/L Irregular menstrual cycles Unilateral ovary Polycystic ovary syndrome Endometriosis Male factor of infertility requiring ICSI History of recurrent miscarriage Endocrinologic disorders Systemic disease contraindicating pregnancy

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 106 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | Three weeks after start of ovarian stimulation
  Oocytes aspirated during ovum pickup

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof, Study Chair — Cairo University; Usama M Fouda, Prof, Study Chair — Riyadh Fertility and Reproductive Health center
Locations (2):
- Egypt (2):
  - Obstetrics &Gynecology Department , Faculty of medicine ,Cairo university, Cairo
  - Riyadh Fertility and Reproductive Health center, Giza

REFERENCES:
- [Background] Badawy A, Mosbah A, Tharwat A, Eid M. Extended letrozole therapy for ovulation induction in clomiphene-resistant women with polycystic ovary syndrome: a novel protocol. Fertil Steril. 2009 Jul;92(1):236-9. doi: 10.1016/j.fertnstert.2008.04.065. Epub 2008 Aug 15. PMID 18706549